CLINICAL TRIAL: NCT07187544
Title: Effect of Co-administration of Carbetocin and Calcium Chloride on Uterine Tone in Patients Undergoing Elective Cesarean Delivery: a Double-blind Randomized Control Trial
Brief Title: Effect of Co-administration of Carbetocin and Calcium Chloride on Uterine Tone in Patients Undergoing Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-02; 300140 (Other: Health Canada)
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage (Primary)
Keywords: calcium; carbetocin; cesarean
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Calcium Chloride; carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium (Active Comparator): Intravenous calcium chloride 10% (1g) will be administered in 100ml normal saline, over 10 minutes.
  Interventions: Drug: Calcium Chloride; Drug: Carbetocin
- Placebo (Placebo Comparator): Intravenous administration of 100ml normal saline, over 10 minutes.
  Interventions: Other: Placebo; Drug: Carbetocin

INTERVENTIONS:
Drug: Calcium Chloride — Intravenous calcium chloride 10% (1g) will be administered in 100ml normal saline, over 10 minutes.
  Arms: Calcium
Other: Placebo — Intravenous administration of 100ml normal saline, over 10 minutes.
  Arms: Placebo
Drug: Carbetocin — 50 mcg intravenous carbetocin.

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal mortality, and its severity has been increasing globally, including in high-income countries. The most common cause of PPH is uterine atony occurring in about 70% of cases. Uterotonic agents, like oxytocin, are key in managing the third stage of labour to prevent PPH. Oxytocin is a short-acting medication and requires frequent dosing, however, carbetocin, a longer-acting analogue that can be administered as a single dose, provides sustained uterotonic activity. Calcium chloride is a readily available, inexpensive medication that has been studied as an adjunct to primary uterotonics due to its role in uterine contractility. A randomized trial found no overall reduction in blood loss with calcium chloride and oxytocin, but a subgroup analysis suggested it may reduce bleeding in cases of uterine atony. This study was conducted in the US where carbetocin is not readily available. The investigators propose a double-blind randomized trial investigating if co-administering calcium chloride with carbetocin during scheduled cesarean deliveries reduces PPH secondary to uterine atony.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled CD for patients ≥ 37 weeks excluding high risk factors for uterine atony
2. Neuraxial anesthesia as the primary anesthetic where intrathecal medications are the primary anesthetic

Exclusion Criteria:

1. Risk factors for uterine atony including:

   1. Overdistended uterus due to fetal macrosomia reported on prenatal ultrasound >90th centile or > 4000 gm, multiple gestation, grand multiparity (≥5 births at ≥ 20 weeks gestation), polyhydramnios
   2. History of uterine atony/PPH (documented with blood loss > 2000 ml, blood transfusion, use of surgical methods such as Bakri balloon, B-Lynch sutures, uterine artery ligation or embolization)
   3. Obesity with body mass index (BMI) > 40 kg/m2
   4. Placenta previa and/or placenta accreta
2. Digoxin therapy within 14 days (hypercalcemia can exacerbate digoxin toxicity)
3. Patients needing intraoperative IV ceftriaxone or tetracycline.
4. Kidney disease including Stage 3 chronic kidney disease, serum creatinine above 120 mmol/L or GFR <60 ml/min (to prevent hypercalcemia due to reduced creatinine clearance in those with impaired kidney function as calcium is renally excreted)
5. Calcium channel blockade within 24 hours (opposing effect)
6. Known history of cardiac disease including arrhythmias, ischemia, and congenital heart disease (to avoid attributing cardiac symptoms to study drugs)
7. Preexisting hypertension, preeclampsia or persistent elevated blood pressure above 160/100 mmHg requiring treatment
8. Emergency cesarean deliveries or women in labor
9. Planned general anesthetic for patients where neuraxial is contraindicated.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Uterine Tone 10 minutes | 10 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 10 minutes post-fetal delivery, utilizing a verbal numeric rating scale of 0-10.

SECONDARY OUTCOMES:
Uterine Tone baseline | 1 minute
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician after delivery of the placenta, utilizing a verbal numeric rating scale of 0-10.
Uterine Tone 5 minutes | 5 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 10 minutes post-fetal delivery, utilizing a verbal numeric rating scale of 0-10.
Uterine Tone 15 minutes | 15 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 15 minutes post-fetal delivery, utilizing a verbal numeric rating scale of 0-10.
Uterine Tone 20 minutes | 20 minutes
  The intensity of uterine tone as evaluated by palpation of the uterus by the obstetrician at 20 minutes post-fetal delivery, utilizing a verbal numeric rating scale of 0-10.
Additional uterotonic agents required intraoperatively | 90 minutes
  The number of patients who are administered additional uterotonic agents intraoperatively will be recorded
Additional uterotonic agents required post-operatively | 24 hours
  The number of patients who are administered additional uterotonic agents post-operatively will be recorded
Semi-quantitative blood loss (SQBL) | 90 minutes
  Blood loss measured in the operating room by volume (ml)
Incidence of postpartum hemorrhage | 24 hours
  The number of patients with blood loss greater than or equal to 1000ml
Presence of blood transfusion | 24 hours
  Number of units of blood product administered post-delivery
Number of patients with conservative surgical methods to manage post partum hemorrhage | 2 hours
  Bakri balloon/B-Lynch sutures used intraoperatively
Number of patients with radiological methods used to manage post partum hemorrhage | 2 hours
  Uterine artery embolization used intraoperatively.
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24 hours | 24 hours
  ObsQoR-10 score at 24 hours. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.
Number of patients with hypotension defined as systolic blood pressure less than 80% of baseline | 2 hours
  Systolic blood pressure < 80% of baseline, at any time during surgeryTime
Number of patients with hypertension defined as systolic blood pressure greater than 120% of baseline | 2 hours
  Systolic blood pressure > 120% of baseline, at any time during surgery
Number of patients with tachycardia defined as heart rate greater than 130% of baseline | 2 hours
  Heart rate > 130% of baseline, at any time during surgery
Number of patients with bradycardia defined as heart rate less than 70% of baseline | 2 hours
  Heart rate < 70% of baseline, at any time during surgery
Presence of atrial fibrillation: ECG | 2 hours
  Presence of atrial fibrillation as recorded by ECG, at any time during surgery
Presence of atrial flutter: ECG | 2 hours
  Presence of atrial flutter as recorded by ECG, at any time during surgery
Presence of nausea: questionnaire | 2 hours
  The presence of nausea at any time during surgery, as reported by the patient
Presence of vomiting: questionnaire | 2 hours
  The presence of vomiting at any time during surgery, as reported by the patient
Number of patients with chest pain: questionnaire | 2 hours
  Any presence of chest pain, at any time during surgery, as reported by the patient
Number of patients with irritation at the intravenous site: questionnaire | 2 hours
  Any presence of irritation, including pain or burning, at the intravenous site, at any time during surgery, as reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No